CLINICAL TRIAL: NCT02767830
Title: Adherence to a Running and Nutrition Program in Children Aged 8-12 Years: A Pilot Study
Brief Title: Cleveland Kids Run
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHCaseMC 2
Record Dates: First submitted 2016-05-08; First posted 2016-05-10 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

ARMS (1):
- Excercise and Nutrition Program (Experimental): Children and their care givers will receive 5 lectures on nutrition and exercise and will be given a weekly running program. At the end of the study children will be encouraged to participate in an annual 0.25-0.5 mile race.
  Interventions: Behavioral: Excercise and Nutrition Program

INTERVENTIONS:
Behavioral: Excercise and Nutrition Program

SUMMARY:
A 12 month long program focused on making good food choices and exercise directed at 8-12 year olds and their caregivers. The program will consist of monthly educational meetings each teaching a new nutritional and exercise concept. Children will be given weekly exercise schedules and their adherence to the program will be assessed. The study will culminate with an annual children's race in May.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 8-12 years old and enrolled in kindergarten through 6th grade in a Cleveland Public School
* Participants must have at least a B-average or equivalent in the prior academic year
* Participants must have at least one part or guardian who is able to accompany the participant during exercise and educational sessions
* Participants must be willing to participate in the Rite Aid Cleveland Marathon Ringling Bros. and Barnum & Bailey Red Nose Run® at the end of the study

Exclusion Criteria:

* Children who are younger than 8 years or older than 12 years

  * Children whose parents who are unable or unwilling to provide informed consent,
  * Children whose parents are are illiterate or non-English speaking or reading
  * Children whose parents are unable or unwilling to accompany them to educational and exercise sessions
  * Children with a medical condition that prevents them from unmonitored exercise
  * Children who have not maintained an equivalent of a B-average in the prior academic year

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to program | 12 months
  number of subjects who participate in race